CLINICAL TRIAL: NCT05938062
Title: Is the Use of Fibrinogen in Cesarean Section Related to Bleeding and Blood Product in Patients With Placenta Accreta Spectrum?: a Retrospective Randomized Study
Brief Title: Fibrinogen Concentrate and Placenta Acreta Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-02
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Obstetric Anesthesia Problems; Placenta Accreta
Keywords: fibrinogen concentrate; obstetric anesthesia; plasenta acreata spectrum; postpartum hemorrhage
MeSH Terms: conditions — Placenta Accreta; Postpartum Hemorrhage | interventions — Fibrinogen

STUDY DESIGN:
Intervention Model Description: retrospective randomized study
Masking Description: retrospective randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- grup 1: the group without fibrinogen concentrate (GNF) (Experimental): grup 1: the group without fibrinogen concentrate (GNF)
  Interventions: Procedure: the group without fibrinogen concentrate (GNF) , the group with fibrinogen concentrate (GF)
- Grup 2: the group with fibrinogen concentrate (Experimental): Grup 2: the group with fibrinogen concentrate
  Interventions: Procedure: the group without fibrinogen concentrate (GNF) , the group with fibrinogen concentrate (GF)

INTERVENTIONS:
Procedure: the group without fibrinogen concentrate (GNF) , the group with fibrinogen concentrate (GF) — the group without fibrinogen concentrate (GNF, ) the group with fibrinogen concentrate (GF)
  Other Names: group 1: the group without fibrinogen concentrate (GNF); group 2: the group with fibrinogen concentrate (GF)

SUMMARY:
The aim of this study is to evaluate the relationship between fibrinogen use and bleeding in patients who underwent cesarean section with a prediagnosis of PAS.

The key question(s) it aims to answer are:

[Does the use of fibrinogen concentrate reduce bleeding in PAS patients?] Patients who had a cesarean section with a pre-diagnosis of PAS were analyzed retrospectively. The choice of anesthesia applied to the patients and the relationship between the use of blood products and bleeding were evaluated.

DETAILED DESCRIPTION:
Our study was designed as a retrospective randomized study. Patients aged 20-50 years and >34 weeks of gestation who accepted the birth with a cesarean section with a pre-diagnosis of PAS were evaluated retrospectively.

examined. were randomized into 2 groups, 53 patients in each group: group1: GNF : the group without fibrinogen concentrate

Group 2: GF: the group with fibrinogen concentrate

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years PAS pre-diagnosed pregnant women
* >34 weeks of pregnancy
* Those with normal renal functions

Exclusion Criteria:

* Patients with renal insufficiency
* Those with <34 weeks of gestation
* Pregnant women with missing data

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 146 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Laboratory hemoglobin level(g/dl) | Change from preoperative to postoperative day 1(POD 1) hemoglobin values (g/dl).
  Our primary aim was to evaluate the postoperative day 1(POD 1) hemoglobin values(g/dl).

SECONDARY OUTCOMES:
The intensive care unit (ICU) admission and length of stay. | postoperatively up to 1 months
  The secondary aim was to investigate the intensive care unit (ICU) admission and length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Akyol, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Duygu Akyol, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morlando M, Collins S. Placenta Accreta Spectrum Disorders: Challenges, Risks, and Management Strategies. Int J Womens Health. 2020 Nov 10;12:1033-1045. doi: 10.2147/IJWH.S224191. eCollection 2020. PMID 33204176
- [Background] Shainker S, Shamshirsaz A, Haviland M, O'Brien K, Redhunt A, Bateni Z, Moaddab A, Fox K, Hui SK, Belfort M, Dildy G, Hacker M. Utilization and outcomes of massive transfusion protocols in women with and without invasive placentation. J Matern Fetal Neonatal Med. 2020 Nov;33(21):3614-3618. doi: 10.1080/14767058.2019.1581168. Epub 2019 Mar 1. PMID 30821559
- [Result] DeSimone RA, Leung WK, Schwartz J. Transfusion Medicine in a Multidisciplinary Approach to Morbidly Adherent Placenta: Preparing for and Preventing the Worst. Transfus Med Rev. 2018 Oct;32(4):244-248. doi: 10.1016/j.tmrv.2018.05.007. Epub 2018 Jun 27. PMID 30025661